CLINICAL TRIAL: NCT06470607
Title: Biological Observational Monocentric Study Aimed at Analyzing the Lymphocytic Infiltrate of Lung Tumors
Brief Title: The Lymphocytic Infiltrate of Lung Tumors.
Acronym: TREGILC
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Pierluigi Novellis, MD, Scientific Institute San Raffaele
Other Study IDs: 117/INT/2022
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Immune System
Keywords: thoracic tumors; Immune checkpoints; lymphocytes
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples include: peripheral blood and tumor tissue. The following will be analyzed: Number of infiltrating lymphocytes; expression of markers of the immune response,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is configured as a monocentric observational transversal biological study.

The main objective of the study is the reconstruction of the molecular organization of tumors of the thoracic cavity, in particular non-small cell lung cancer (NSCLC).

The study involves the collection of clinical data and biological material (blood and tumor tissue) from 70 subjects diagnosed with thoracic tumors.

DETAILED DESCRIPTION:
Inclusion criteria:

The study population will include all patients with the following characteristics:

* Ability to provide informed consent
* Men and women over the age of 18 years old
* Patients candidates for surgical treatment diagnosed with thoracic tumors

The procedures to which the patient will undergo during the study follow the standard of clinical practice for the treatment of pathology.

Exclusion criteria:

* Previous chemotherapy for any cancer within the last 6 months
* Pregnant and/or breastfeeding women
* Immunosuppressive state (states of immunosuppression or ongoing immunosuppressive/immunomodulatory treatments)

The time of observation of the patient for the purposes of the study is limited to the time of hospitalization and the surgical procedure, the patient will therefore perform a single visit to the hospital and there is no provision for the collection of further data following discharge. The study involves a single timepoint of data collection and samples.

The study will have a total duration of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent;
* Men and women over the age of 18;
* Patients candidates for surgical treatment diagnosed with thoracic tumors

Exclusion Criteria:

* Previous chemotherapy for any cancer within the last 6 months;
* Pregnant and/or breastfeeding women;
* Immunosuppressive state (states of immunosuppression or ongoing immunosuppressive/immunomodulatory treatments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is made up of patients diagnosed with thoracic cancer, candidates for surgical resection for the disease.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
LYMPHOCYTE ISOLATION | from enrollment in the study to surgery at 15 days
  the collection of lymphocytes, and their sequencing and analysis of differentially expressed genes.

SECONDARY OUTCOMES:
Lymphocyte gene expression | from surgery to processing within 48 hours
  Analysis of gene expression and translational activity of lymphocyte cells (CD4+)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute Ospedale San Raffaele, Milan, Italy